CLINICAL TRIAL: NCT06139250
Title: Development of a High-speed Multimodal Photoacoustic/Ultrasound System for Functional Imaging of the Neonatal Brain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-brain
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hypoxia-Ischemia, Brain
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypoxic-ischemic encephalopathy group: Photoacoustic/ultrasound imaging will be used for neonates with hypoxic ischemic encephalopathy
- control group: Photoacoustic/ultrasound imaging will be used for neonates without brain disease

SUMMARY:
In today's medical field, there is a growing emphasis on the development of functional and molecular imaging. Therefore, it has significant technical limitations.

To address this issue, this project aims to develop a high-speed multimodal photoacoustic/ultrasound functional imaging system that provides both structural and functional information of tissue and organs, thus enhancing the accuracy of early screening and diagnosis of neonatal cranial lesions. This imaging technology is entirely non-invasive and does not involve ionizing radiation or contrast agents. Products using the same technology have already received FDA approval and entered clinical use in the United States. We develop a new generation of multimodal photoacoustic/ultrasound functional imaging equipment to reveal the physiological characteristics and structural details of neonatal cranial lesions, offering advantages and complementary information compared to traditional medical imaging methods.

DETAILED DESCRIPTION:
Medical imaging plays a huge role in clinical diagnosis. At present, the commonly used imaging methods for neonatal brain imaging include ultrasound imaging, magnetic resonance imaging, and CT. Due to the imaging scale, speed, and radiation limitation, large imaging devices such as CT and magnetic resonance imaging usually have limitations in the early screening and diagnosis of neonatal brain lesions. With the advantages of flexibility and convenience, ultrasound has become a common imaging method for neonatal brain organs. However, conventional ultrasound imaging usually only provides structure-related information, and it is difficult to reveal the physiological characteristics of the lesions. Therefore, this project aims to develop a high-speed multi-modal photoacoustic/ultrasound functional imaging system to provide structural and functional information of tissues and organs, thereby improving the accuracy of early screening and diagnosis of neonatal brain lesions. The imaging technique is completely noninvasive and does not use any ionizing radiation or contrast media. A product that uses the same technology as this imaging device has been approved by the FDA and entered the clinic in the United States.

The imaging device consists of two imaging modalities, photoacoustic imaging and ultrasound imaging. Photoacoustic imaging (PAI) can be used to image the optical absorption characteristics of human tissues by safely irradiating the human body with near-infrared light (complying with international safety standards) to produce a short time temperature rise (less than 0.1 degrees Celsius), resulting in a weak ultrasound signal. The ultrasonic imaging principle of the device is the same as that of clinical B-ultrasound, which uses ultrasound to safely irradiate the body (obeying international safety standards) and obtain reflected signals. This project is supported by the Young Scientist Project of Diagnosis and Treatment Equipment of the Key Research and Development Program of the Ministry of Science and Technology, jointly applied by the research group of Teacher Lin Li from Zhejiang University and the research group of Huang Pin from the Second Affiliated Hospital of Zhejiang University School of Medicine. This project aims to develop a new generation of multimodal photoacoustic/ultrasound functional imaging equipment to reveal the physiological characteristics and structural details of neonatal brain lesions. And traditional medical imaging methods form advantages and information complementary.

ELIGIBILITY:
Inclusion Criteria:

① All patients were clinically diagnosed as hypoxic-ischemic encephalopathy. ② infants born within 1-7 days (including 7 days); ③ The gestational age was 37-42 weeks; ④ body weight between 2.5kg and 4kg; ⑤ Color Doppler ultrasound and magnetic resonance imaging were performed in all patients. ⑥ Complete clinical records

Exclusion Criteria:

① Children with contraindications to MRI examination; ② Brain tumor, congenital heart disease; ③ unclear clinical diagnosis; ④ a definite history of intrauterine infection; ⑤ image quality affects the diagnosis of newborns; ⑥ Lack of complete clinical medical records.

Ages: 1 Day to 7 Days | Sex: All
Age Groups: Child
Study Population: 1. Neonates with hypoxic ischemia encephalopathy group ① All patients were clinically diagnosed as HIE. ② infants born within 1-7 days (including 7 days); ③ The gestational age was 37-42 weeks; ④ body weight between 2.5kg and 4kg; ⑤ Color Doppler ultrasound and magnetic resonance imaging were performed in all patients. ⑥ Complete clinical records
  2. Control group：① There was no neonatal encephalopathy. ② born within 1-7 days (including 7 days); ③ The gestational age was 37-42 weeks; ④ Body weight between 2.5kg and 4kg
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy | one year
  The photoacoustic/ultrasound multimodal functional imaging data can be used to analyze the specific physiological characteristics of neonatal brain lesions and evaluate the diagnostic basis. The expected accuracy of this technology in diagnosing specific brain lesions can be evaluated before the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pintong Huang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Department of Ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal